CLINICAL TRIAL: NCT00001584
Title: Determination of HIV-1 Production by the Prostate
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970158; 97-C-0158
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-05

CONDITIONS: HIV Infections
Keywords: Pathogenesis; Resistance; Sanctuary Sites; Semen; Sexual Transmission
MeSH Terms: conditions — HIV Infections

SUMMARY:
Virus present in semen likely contributes substantially to the sexual transmission of HIV. However, the source of HIV in semen is unknown. Some evidence suggests that the prostate may be the source of at least some of the virus in semen. This study is designed to determine whether the prostate may serve as the source of virus in semen by comparing the concentration of HIV-1 RNA in semen donated normally, in semen obtained following prostatic massage, and in expressed prostatic secretions. Finding a source for semen HIV would provide important insights into several aspects of HIV sexual transmission. Since some drugs do not enter the prostate well, the finding that virus is produced in the prostate might suggest the prostate could serve as a reservoir for HIV, leading to the development of resistance to antiviral agents.

DETAILED DESCRIPTION:
Virus present in semen likely contributes substantially to the sexual transmission of HIV. However, the source of HIV in semen is unknown. Some evidence suggests that the prostate may be the source of at least some of the virus in semen. This study is designed to determine whether the prostate may serve as the source of virus in semen by comparing the concentration of HIV-1 RNA in semen donated normally, in semen obtained following prostatic massage, and in expressed prostatic secretions. Finding a source for semen HIV would provide important insights into several aspects of HIV sexual transmission. Since some drugs do not enter the prostate well, the finding that virus is produced in the prostate might suggest the prostate could serve as a reservoir for HIV, leading to the development of resistance to antiviral agents.

ELIGIBILITY:
HIV positive male.

Willing and able to participate on study.

Age greater than or equal to 18 years.

Stable antiretroviral therapy for the preceding 4 weeks and judged likely to remain on stable therapy for the study.

Patients with a history of vasectomy or orchiectomy may be admitted to the study, but the data obtained from those patients will be analyzed separately on a pilot basis.

Able to provide informed consent.

Clinically stable.

No clinical or laboratory evidence of bacterial prostatitis.

No clinical or laboratory evidence of genito-urinary tract infection.

No history of prostatectomy.

Absolute neutrophil count greater than 500/ul.

Platelets greater than 50,000.

Patient must not have had treatment within the prior 8 weeks with anti-androgens or estrogens. Stable therapy with anabolic steroids will be allowed.

Patient must not have localized or systemic disease which would, in the opinion of the investigator(s), render the patient at risk following prostatic massage and/or the donation of semen.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 1997-07; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hamed KA, Winters MA, Holodniy M, Katzenstein DA, Merigan TC. Detection of human immunodeficiency virus type 1 in semen: effects of disease stage and nucleoside therapy. J Infect Dis. 1993 Apr;167(4):798-802. doi: 10.1093/infdis/167.4.798. PMID 8450243
- [Background] Liuzzi G, Chirianni A, Clementi M, Bagnarelli P, Valenza A, Cataldo PT, Piazza M. Analysis of HIV-1 load in blood, semen and saliva: evidence for different viral compartments in a cross-sectional and longitudinal study. AIDS. 1996 Dec;10(14):F51-6. doi: 10.1097/00002030-199612000-00001. PMID 8970677
- [Background] Van Voorhis BJ, Martinez A, Mayer K, Anderson DJ. Detection of human immunodeficiency virus type 1 in semen from seropositive men using culture and polymerase chain reaction deoxyribonucleic acid amplification techniques. Fertil Steril. 1991 Mar;55(3):588-94. PMID 2001759